CLINICAL TRIAL: NCT04371900
Title: The Effects of Unintended Pregnancy on Children
Brief Title: Michigan Contraceptive Access, Research, and Evaluation Study Children: Phase 1
Acronym: M-CARES-K
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: Planned Parenthood Federation of America (Other); National Opinion Research Center (Other)
Responsible Party: Principal Investigator, Martha Bailey, Adjunct Research Professor, Population Studies Center, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: HUM00132909B
Record Dates: First submitted 2020-04-29; First posted 2020-05-01 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy
Keywords: contraception; financial access to reproductive health care; unintended pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Experimental Group (Experimental): Mothers randomized to receive a voucher to be used at Planned Parenthood to cover the cost of contraceptives
  Interventions: Behavioral: Mother receives voucher valued at 100% of cost of name-brand IUD (March 4, 2019-March 31, 2023); Behavioral: Mother receives voucher valued at 50% of cost of name-brand IUD (August 26, 2018-March 3, 2019)
- Control Group (No Intervention): Mothers randomized to NOT receive a voucher. Mothers in this arm receive the Planned Parenthood standard of care priced according to the Planned Parenthood sliding scale.

INTERVENTIONS:
Behavioral: Mother receives voucher valued at 100% of cost of name-brand IUD (March 4, 2019-March 31, 2023) — M-CARES randomized vouchers for contraception valued up to 100% of inserting a name-brand IUD (e.g., Skyla, Paraguard, Mirena) for women with out of pocket costs at Planned Parenthood. This intervention occurred from March 4, 2019, forward.
  Arms: Experimental Group
Behavioral: Mother receives voucher valued at 50% of cost of name-brand IUD (August 26, 2018-March 3, 2019) — M-CARES randomized vouchers for contraception valued up to 50% of inserting a name-brand IUD (e.g., Skyla, Paraguard, Mirena) for women with out of pocket costs at Planned Parenthood. This intervention occurred after November 4, 2019.
  Arms: Experimental Group

SUMMARY:
This project builds on the Michigan Contraceptive Access Research and Evaluation Study (M-CARES) to evaluate the long-term effects of mothers' access to free contraceptives and reductions in unintended pregnancies on their children's well-being.

DETAILED DESCRIPTION:
M-CARES uses a randomized control trial design to assess the effects of providing free contraception to mothers on their children born before the intervention. The population subject to intervention is fecund women age 18-35 years at risk of pregnancy and who are clients at Planned Parenthood clinics of Michigan (PPMI), who meet income eligibility criteria, and who would otherwise pay out-of-pocket for services on the day of recruitment (i.e., lacking insurance coverage for received service). The experimental (treatment) condition is a mother's receipt of a voucher providing access to no-cost contraception (up to the price of a name-brand intrauterine device) for 100 days. The control group of mothers receives no voucher. All enrolled women complete a two-part baseline survey and consent to be re-contacted for two follow-up interviews in outgoing years. They also complete a two-part baseline survey and consent to be re-contacted for two follow up interviews in outgoing years. In addition, mothers consent to linkages to their own and their children's administrative data from records held by state and federal health, education, criminal justice, and tax records. Consent covers children already born to women at the time of intervention and children born after intervention. Survey and administrative data provide outcome measures to assess children's well-being and development up to age 18. The study will compare children of mothers who receive the intervention to those who did not.

ELIGIBILITY:
Inclusion Criteria:

The proposed project will analyze the outcomes of children ages 0 to 17 years old whose mothers enrolled in the Michigan Contraceptive Access, Research and Evaluation Study (M-CARES). M-CARES participation requires that mothers are:

* 18-35 years old
* physically capable (biologically female and fecund) and at risk of having a pregnancy,
* not pregnant at the time of enrollment
* not wishing to become pregnant in the 12 months after enrollment,
* are seeking care at Planned Parenthood of Michigan, and
* face out-of-pocket costs for contraceptives at Planned Parenthood of Michigan.

Ages: 0 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4700 (Estimated)
Dates: Start 2018-08-26 (Actual); Primary Completion 2049-12-31 (Estimated); Study Completion 2049-12-31 (Estimated)

PRIMARY OUTCOMES:
Number of siblings born after study enrollment (1 year) | Up to 1 year post enrollment
  Number of children born to individual's mother as determined in mother's survey responses and Vital Records (count: 0, 1, 2....)
Number of siblings born after study enrollment (3 year) | Up to 3 year post enrollment
  Number of children born to individual's mother as determined in mother's survey responses and Vital Records (count: 0, 1, 2....)
Number of siblings born after study enrollment (5 year) | Up to 5 year post enrollment
  Number of children born to individual's mother as determined in mother's survey responses and Vital Records (count: 0, 1, 2....)
Standardized achievement test score (1 year) | Up to 1 year post enrollment
  Percentile on state standardized achievement test (range: 1-100)
Standardized achievement test score (3 year) | Up to 3 year post enrollment
  Percentile on state standardized achievement test (range: 1-100)
Standardized achievement test score (5 year) | Up to 5 year post enrollment
  Percentile on state standardized achievement test (range: 1-100)

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - Planned Parenthood - Ann Arbor-West, Ann Arbor, Michigan
  - Planned Parenthood - Detroit, Detroit, Michigan
  - Planned Parenthood - Ferndale, Ferndale, Michigan
  - Planned Parenthood - Grand Rapids, Grand Rapids, Michigan
  - Planned Parenthood - Kalamazoo, Kalamazoo, Michigan
  - Planned Parenthood - Lansing, Lansing, Michigan
  - Planned Parenthood - Livonia, Livonia, Michigan
  - Planned Parenthood - Traverse City, Traverse City, Michigan
  - Planned Parenthood - Warren, Warren, Michigan

IPD SHARING:
Plan to Share IPD: No